CLINICAL TRIAL: NCT00513500
Title: Zambia Integrated Management of Malaria and Pneumonia Study
Acronym: ZIMMAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Center for International Health and Development (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Kojo Yeboah-Antwi, Center for International Health and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GHS-A-00-00020-00-5
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Results first posted 2010-07-13 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Pneumonia; Malaria
Keywords: community health care; community health worker; malaria; pneumonia; rapid diagnostic test
MeSH Terms: conditions — Pneumonia; Malaria | interventions — Artemether, Lumefantrine Drug Combination; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Give one half tablet (20mg artemether, 120mg lumefantrine) to children weighing (5-9.9kg) and one tablet to children weighing (10-20kg) twice a day for three days for malaria based on rapid diagnostic test. For pneumonia, give one half tablet (250mg amoxicillin) for children weighing (5-9.9kg) and one tablet for children weighing (10-20kg) three times a day for five days.
  Interventions: Drug: Coartem and amoxicillin
- 2 (Active Comparator): Give one half tablet (20mg artemether, 120mg lumefantrine) to children weighing (5-9.9kg) and one tablet to children weighing (10-20kg) twice a day for three days for malaria based on clinical diagnosis. For pneumonia, refer to the nearest health facility
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: Coartem and amoxicillin — Perform RDT and give Coartem for malaria and give amoxicillin for fast breathing
  Arms: 1
Drug: Coartem — Give Coartem without RDT and refer fast breathing
  Arms: 2

SUMMARY:
The purpose of the study is to demonstrate the effectiveness and feasibility of community-based management of pneumonia and malaria by community health workers (CHWs) in a rural district of Zambia.

DETAILED DESCRIPTION:
Pneumonia and malaria are the two leading causes of morbidity and mortality among children under five in sub-Saharan Africa. Due to limited access to health services in many developing countries, a number of global health organizations, including the World Health Organization, have strongly advocated the use of community health workers (CHWs) to deliver basic health care in the community and to facilitate referral to primary health facilities.

Existing supported CHWs in the study area will be trained in the assessment and classification of children between six months and five years of age presenting with fever and/or cough/difficult breathing. In the intervention arm, CHWs will be supplied with rapid diagnostic tests (RDTs), Coartem (a fixed dose combination of artemether-lumefantrine) and amoxicillin. The intervention CHWs will be trained to use RDTs in patients with reported fever and provide those with a positive result with Coartem; and patients suspected of pneumonia (based on fast breathing) will be treated with amoxicillin as per the standard of care at health facilities and monitored. In the control arm, no RDT will be performed. The CHWs will be supplied with Coartem to treat malaria/febrile illness as per the integrated management of childhood illnesses (IMCI) guidelines and patients suspected of pneumonia will be referred to the health facility for treatment as per the current practice. Data collectors will routinely visit CHWs to collect data on their consultations and follow-up patients treated by CHWs in their homes..

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months and 5 years
* Present with history of fever or reported fever
* Present with cough or difficult breathing

Exclusion Criteria:

* Age below 6 months and above 5 years
* Presence of signs and symptoms of severe illness

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3125 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kojo Yeboah-Antwi, MD, MPH, Principal Investigator — Center for International Health and Development
Locations (1):
- Chikankata Health Services, Chikankata, Southern Province, Zambia

REFERENCES:
- [Derived] Yeboah-Antwi K, Pilingana P, Macleod WB, Semrau K, Siazeele K, Kalesha P, Hamainza B, Seidenberg P, Mazimba A, Sabin L, Kamholz K, Thea DM, Hamer DH. Community case management of fever due to malaria and pneumonia in children under five in Zambia: a cluster randomized controlled trial. PLoS Med. 2010 Sep 21;7(9):e1000340. doi: 10.1371/journal.pmed.1000340. PMID 20877714

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Treatment: Intervention: Treatment for malaria and pneumonia:
  Treat malaria based on rapid diagnostic test with half tablet (20mg artemether, 120mg lumefantrine) for children weighing 5-9.9kg and one tablet (20mg artemether, 120mg lumefantrine) for children weighing 10-20kg twice a day for three days.
  Treat pneumonia with half tablet (250mg amoxicillin) for children weighing 5 - 9.9kg and one tablet (250mg amoxicillin for children weighing 10-20kg three times a day for five days.
- Current Practice: Control: Treatment for malaria and pneumonia referral Treat malaria based on fever with half tablet (20mg artemether, 120mg lumefantrine) for children weighing 5-9.9kg and one tablet (20mg artemether, 120mg lumefantrine) for children weighing 10-20kg twice a day for three days.
  Refer children with pneumonia to the nearest health facility.
Period: Overall Study
Arm/Group | Enhanced Treatment | Current Practice
Started | 1017 | 2108
Completed | 976 | 2054
Not Completed | 41 | 54
Not completed — Lost to Follow-up | 35 | 39
Not completed — Death | 2 | 1
Not completed — Hospitalized | 4 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Treatment | Current Practice | Total
Number analyzed (Participants) | 1017 | 2108 | 3125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1017 | 2108 | 3125
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: months] | 22.6 (14.0) | 23.6 (14.7) | 23.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 484 | 1028 | 1512
  Male | 533 | 1080 | 1613
Region of Enrollment [Number; unit: participants]
  Zambia | 1017 | 2108 | 3125

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Who Received Early and Appropriate Treatment for Pneumonia.
Description: Early and appropriate is defined as receiving 13-15 doses of amoxicillin over 5 days and receiving the first dose within 24-48 hours of onset of first symptom
Time Frame: one year
Population: The number of participants determined for this analysis was based on those classified as pneumonia. The analysis was based on an intent-to-treat basis.
Measure: Number; unit: partcipants
Arm/Group | Enhanced Treatment | Current Practice
Number analyzed (Participants) | 362 | 203
partcipants | 247 | 27
Statistical Analysis 1: Comparison: Enhanced Treatment vs Current Practice; Test type: Superiority or Other; Risk Ratio (RR) = 5.32, 95% CI [2.19 to 8.94]

2. Primary Outcome: Number of Children With Fever Who Received Coartem (Artemether-lumefantrine)
Time Frame: one year
Population: The participants analyzed was based on children reported with fever. Analysis was per intention to treat.
Measure: Number; unit: participants
Arm/Group | Enhanced Treatment | Current Practice
Number analyzed (Participants) | 963 | 2084
participants | 265 | 2066
Statistical Analysis 1: Comparison: Enhanced Treatment vs Current Practice; Test type: Superiority or Other; Risk Ratio (RR) = 0.23, 95% CI [0.14 to 0.38]

3. Secondary Outcome: Number of Children Who do Not Respond to Treatment for Pneumonia
Time Frame: one year
Population: Based on number classified as having pneumonia. Analysis was per intention to treat
Measure: Number; unit: participants
Arm/Group | Enhanced Treatment | Current Practice
Number analyzed (Participants) | 362 | 203
participants | 41 | 41
Statistical Analysis 1: Comparison: Enhanced Treatment vs Current Practice; Test type: Superiority or Other; Risk Ratio (RR) = 0.44, 95% CI [0.21 to 0.93]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patients were followed up on Day 5-7 and caregivers were specifically asked about adverse events and documented on a case report form.
  The participants at risk to RDT related adverse events in the Enhanced Treatment Arm were 973 because RDT was not done on 44 subjects (no fever = 36; refused = 6; and poor light at the time of visit =2).
Arm/Group | Enhanced Treatment | Current Practice
Serious Adverse Events (participants affected / at risk) | 6/1017 | 15/2108
Other Adverse Events (participants affected / at risk) | 16/973 | 0/2018
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Treatment (N=1017) | Current Practice (N=2108)
Deaths (Infections and infestations) | 2 (1017) | 1 (2108)
Hospitalization (Infections and infestations) | 4 (1017) | 14 (2108)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Treatment (N=973) | Current Practice (N=2018)
RDT related (Skin and subcutaneous tissue disorders) | 16 (16) | 0 (0) — These adverse effects with related to pricking the finger to take blood for rapid diagnostic test

LIMITATIONS AND CAVEATS:
Imbalance in enrollment. More patients enrolled in the control arm possibly due to many control community health workers working full time and available to see patients all day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes